CLINICAL TRIAL: NCT05996965
Title: Evaluation of Clinical Utility of Non-invasive Hemodynamic Monitoring Device (HemoVista™) in the Clinical Filed
Brief Title: Evaluation of Clinical Utility of Non-invasive Hemodynamic Monitoring Device
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Other Study IDs: HemoVista
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: HemoVista — additional attatchment of non-invasive hemodynamic monitoring HemoVista with FloTrac

SUMMARY:
In patients undergoing surgery under general anesthesia, the clinical utility of non-invasive hemodynamic status monitoring equipment using HemoVista is compared with invasive hemodynamic status monitoring equipment FloTrac.

DETAILED DESCRIPTION:
For patients who are scheduled to monitor invasive blood pressure, invasive hemodynamic monitoring using FloTrac and additional HemoVista sensors are attached and output data are obtained at the same time during general anesthesia. FloTrac is used to conduct conventional anesthesia and fluid therapy, and the accuracy of HemoVista, a non-invasive hemodynamic monitoring equipment, is compared through prospective observational studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 20 or older who undergo surgery under general anesthesia for more than two hours
* invasive close hemodynamic monitoring with FloTrac is needed

Exclusion Criteria:

* problems in site where HemoVista is attached

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 20 or older
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
degree of agreement in cardiac output | during surgery
  degree of agreement in cardiac output between HemoVista and FloTrac

CONTACTS AND LOCATIONS:
Locations (1):
- Hee-Soo Kim, Seoul, Soul-t'ukpyolsi, South Korea